CLINICAL TRIAL: NCT03293615
Title: Exercise Capacity of Patients with Dermatomyosisthe Role of Muscle Mitochondria and Reactive Oxygen Species
Brief Title: Exercise Capacity of Patients with Dermatomyosis
Acronym: MIDE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: problèmes de recrutement
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6431
Record Dates: First submitted 2017-09-15; First posted 2017-09-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dermatomyositis
MeSH Terms: conditions — Dermatomyositis | interventions — Space Flight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dermatomyositis (DM) (Experimental): Patients with dermatomyositis according to ENMC criteria
  Interventions: Other: exploration
- Non-dermatomyositis inflammatory myopathies (Active Comparator): Patients with other inflammatory myopathy than dermatomyositis according to ENMC criteria
  Interventions: Other: exploration
- No myopathy (No Intervention): Patients without myopathy on muscle biopsy

INTERVENTIONS:
Other: exploration — Difference of the following parameters in patients i) with DM, ii) with another inflammatory myopathy iii) without neuromuscular disease.
  Arms: Dermatomyositis (DM); Non-dermatomyositis inflammatory myopathies

SUMMARY:
Dermatomyositis (DM) patients experience muscle weakness and low aerobic capacities, which are associated with poor health status and increased mortality. The origin of this muscle impairment remains unknown.

The investigators hypothesize that mitochondria functioning is impaired in DM muscle and links with exercise capacities.

ELIGIBILITY:
Inclusion Criteria:

* Woman or man> 18 years,
* Signature of informed consent,
* Muscle biopsy for suspicion of recent inflammatory myopathy (<6 months) or for exclusion of neuromuscular pathology.

Prospectively, following the results of the muscle biopsy, the subjects will divided into three groups meeting the following criteria:

* "DM" group: DM according to the ENMC criteria;
* "other inflammatory myopathy" group: polymyositis, autoimmune necrotizing myopathy, non-specific myositis or inclusion myositis according to the ENMC criteria;
* Group "no neuromuscular pathology": i) myalgia and / or intolerance to exercise and ii) normal neuromuscular examination, iii) no increase in blood creatine kinase level, iv) absence of electromyographic abnormality, v) histological Muscle mass.

Exclusion Criteria:

* - Taking an immunomodulatory treatment within 6 months before inclusion,
* Paraneoplastic form of the disease,
* Presence of associated interstitial pneumonitis,
* Neuromuscular pathology different from inflammatory myopathy,
* Unbalanced cardiovascular disease,
* Impossibility of giving the subject informed information (subject in an emergency situation, difficulty in understanding the subject, ...),
* Subject under safeguard of justice,
* Subject under tutelage or under curators,
* Pregnancy (positive pregnancy test)
* Breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Difference in the capacity of muscle fibers to consume oxygen in the muscle of patients i) with DM, ii) with other inflammatory myopathy, iii) without neuromuscular disease. | Baseline
  This difference in mitochondrial breathing capacity in the muscle will be achieved by: Muscle biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Alain Meyer, Principal Investigator — Les Hôpitaux Universitaires de Strasbourg
Locations (1):
- Meyer, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No